CLINICAL TRIAL: NCT03277339
Title: Psycho-biological Substrates of Therapeutic Benefit of Thermal Cure on Generalized Anxiety Disorders (Insula-TOP)
Brief Title: Psycho-biological Substrates of Therapeutic Benefit of Thermal Cure on Generalized Anxiety Disorders
Acronym: Insula-TOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Collaborators: Association Francaise pour la Recherche Thermale (Other); Les thermes de Saujon (Unknown); Poitiers University Hospital (Other); Centre National de la Recherche Scientifique (CeRCA, umr 7295), France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: InsulaTOP
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Generalized Anxious Disorders
Keywords: Generalized anxious disorders; Thermal cure; paroxetine
MeSH Terms: interventions — Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paroxetine (Experimental): Paroxetine (Deroxat®) Posology : 20 mg per day for 3 weeks. After 2 weeks of treatments, if indicated, physicians will prescribe until 50 mg.
  Interventions: Drug: Paroxetine
- Thermal cure (Other): This study is controlled with a comparator which is the Thermal cure. Thermal cure is realized for 3 weeks.
  Interventions: Other: Thermal cure

INTERVENTIONS:
Drug: Paroxetine — Deroxat® (20 mg/day) 3 week; can be increase on week 2 until 50 mg.
  Arms: Paroxetine
Other: Thermal cure — Thermal cure is realized for 3 weeks
  Arms: Thermal cure

SUMMARY:
Multicenter study comparing paroxetine (n=30) versus thermal cure (n=30) in patients with a diagnosis of Generalised Anxiety Disorders

DETAILED DESCRIPTION:
Multicenter study comparing paroxetine (n=30) versus thermal cure (n=30) in patients with a diagnosis of Generalised Anxiety Disorders

Main objective is to quantify the therapeutic benefit of a thermal cure on generalized anxiety disorders and to understand the psycho-biological substrates of this improvement.

Secondary objectives:

* A decrease of Insula activity at rest during the answers to aversive pictures and during the task of subjective measurement of heartbeat.
* A decrease of sensibility to emotional interference by subliminal presentation of emotional words thanks to a lexical task and a color recognition task associated to simultaneous measurement of physiological indicator of emotional activity ( dermal resistance)

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of generalized anxiety disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM IV)
* No treatment by antidepressant for at least 2 months
* No treatment by anxiolytic/neuroleptic/bete blockers/antipsychotic for at least 3 weeks
* Global score of Hamilton Anxiety Scale (HAM-A) is greater or equal to 20
* Score of HAM-A symptoms greater or equal to 8
* Score of Hamilton Depressive Scale (HAM-D) lower or equal to 7
* Age: Participants will be males and females, 18-75 years of age included.
* For women, no ongoing pregnancy/ negative pregnancy test
* No wounds
* Affiliation to a social security system (recipient or assignee)
* Signed written inform consent form

Exclusion Criteria:

* Treatment by antidepressant for at least 2 months or a treatment by anxiolytic, neuroleptic for at least 3 weeks
* Psychotropic treatment (antidepressant, anxiolytic and neuroleptic) between the preinclusion and inclusion
* Psychotherapy during the 3 months prior to the inclusion
* Thermal cure during the 6 months prior to the inclusion
* Treatment by paroxetine for at least 1 month with dose equal or superior to 20 mg per day during the 12 months prior to the inclusion
* Contraindication to paroxetine
* Enhanced protection (minors, pregnancies women, nursing women,people deprived of liberty by administrative or judicial decision, ...)
* Blood donation during the 3 months prior to the inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Decrease Insula activity during a resting state task | The evaluation of primary end point is performed between day 1 and day 24

SECONDARY OUTCOMES:
Changes of HAM-A score between day 1 and day 24. | The evaluation of primary end point is performed between day 1 and day 24
Sensibility non conscientious to emotional interference in lexical task and in color identification task | D= Day D1/D24/D56
Modulation of electrodermal response during presentation of predictive stimuli on aversive images and its links to the subjective view of emotional state | D= Day D24
Modulation of electrodermal response during presentation of predictive stimuli on aversive images and insula activation | D= Day D24
Lost of significant correlation (Day 24) between HAM-A score, introspective acuity and insula hyperactivation | D= Day D24
Evolution (Day 1 and Day 24) of the correlation between HAM-A global score and 1- the measure of heartbeat 2- emotional reactivity during aversive images task. | D= Day D1/D24.
Difference (Day 1 and Day 24) of correlations between the symptoms severity and the activation of insula cortex during 1-aversive images task, 2-heartbeat measure task. | D= Day D1/D24.
Evaluation of efficacy of the thermal cure Day 56 using HAM-A score | D= Day D56

CONTACTS AND LOCATIONS:
Overall Officials: JAAFARI Nematollah, MD-PhD, Principal Investigator — Centre Hospitalier Henri Laborit; INGRAND Pierre, MD-PhD-PU-PH, Study Chair — Centre d'investigation clinique INSERM CIC P802
Locations (2):
- France (2):
  - Centre Hospitalier Henri Laborit, Poitiers
  - Les thermes de Saujon, Saujon

REFERENCES:
- [Background] Jaafari N, Rachid F, Rotge JY, Polosan M, El-Hage W, Belin D, Vibert N, Pelissolo A. Safety and efficacy of repetitive transcranial magnetic stimulation in the treatment of obsessive-compulsive disorder: a review. World J Biol Psychiatry. 2012 Mar;13(3):164-77. doi: 10.3109/15622975.2011.575177. Epub 2011 May 30. PMID 21623668
- [Background] Jaafari N, Baup N, Bourdel MC, Olie JP, Rotge JY, Wassouf I, Sharov I, Millet B, Krebs MO. Neurological soft signs in OCD patients with early age at onset, versus patients with schizophrenia and healthy subjects. J Neuropsychiatry Clin Neurosci. 2011 Fall;23(4):409-16. doi: 10.1176/jnp.23.4.jnp409. PMID 22231312
- [Background] Jaafari N, Aouizerate B, Tignol J, El-Hage W, Wassouf I, Guehl D, Bioulac B, Daniel ML, Lacoste J, Gil R, Burbaud P, Rotge JY; Insight Study Group. The relationship between insight and uncertainty in obsessive-compulsive disorder. Psychopathology. 2011;44(4):272-6. doi: 10.1159/000323607. Epub 2011 May 6. PMID 21546788
- [Background] Girard SL, Gauthier J, Noreau A, Xiong L, Zhou S, Jouan L, Dionne-Laporte A, Spiegelman D, Henrion E, Diallo O, Thibodeau P, Bachand I, Bao JY, Tong AH, Lin CH, Millet B, Jaafari N, Joober R, Dion PA, Lok S, Krebs MO, Rouleau GA. Increased exonic de novo mutation rate in individuals with schizophrenia. Nat Genet. 2011 Jul 10;43(9):860-3. doi: 10.1038/ng.886. PMID 21743468
- [Background] Dubois O, Salamon R, Germain C, Poirier MF, Vaugeois C, Banwarth B, Mouaffak F, Galinowski A, Olie JP. Balneotherapy versus paroxetine in the treatment of generalized anxiety disorder. Complement Ther Med. 2010 Feb;18(1):1-7. doi: 10.1016/j.ctim.2009.11.003. Epub 2010 Jan 6. PMID 20178872